CLINICAL TRIAL: NCT06416072
Title: Alzheimer's Plasma Extension
Acronym: APEX
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Alzheimer's Clinical Trials Consortium (ACTC) (Unknown); Alzheimer's Therapeutic Research Institute (Other); Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Paul S. Aisen, Professor, University of Southern California
Other Study IDs: ATRI-013; 5R01AG054029 (NIH)
Record Dates: First submitted 2023-02-21; First posted 2024-05-16 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Preclinical Alzheimer's Disease; Early Preclinical Alzheimer's Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group A: Approximately 500 participants who screen failed from the AHEAD study that were plasma positive / PET negative
- Group B: Approximately 250 participants who screen failed from the AHEAD study that were plasma negative / PET negative
- Group C: Approximately 250 participants who screen failed prior to PET imaging will undergo amyloid PET imaging with NAV4694 injection.
  Interventions: Radiation: NAV4694

INTERVENTIONS:
Radiation: NAV4694 — Amyloid PET imaging with NAV4694 injection
  Other Names: [18F]NAV4694
  Groups: Group C

SUMMARY:
The APEX study is a multicenter, observational study designed to capture longitudinal follow-up of plasma biomarkers and cognitive and functional assessments on individuals who screen failed in the AHEAD study over approximately 4 years.

Approximately 1000 participants will be enrolled across three groups:

* Group A: Approximately 500 participants who are discordant on screening (plasma positive / Positron Emission Tomography (PET) negative),
* Group B: Approximately 250 participants who are concordant on screening (plasma negative / PET negative), and
* Group C: Approximately 250 participants selected from the individuals who previously screen failed prior to PET for the AHEAD study with oversampling of racial and ethnic populations underrepresented in Alzheimer's disease (AD) clinical trials.

Primary Objectives:

* Collect longitudinal cognitive and functional assessments and blood-based biomarker data
* Evaluate, characterize, and compare the longitudinal cognitive and functional data between the three groups of participants
* Compare longitudinal change across race and ethnicity, sex, and Apolipoprotein E (ApoE) status

Exploratory Objectives:

• Collect baseline amyloid PET on participants without prior amyloid PET data (Group C)

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of the participant's informed consent to study procedures and for the use of protected health information (HIPAA Authorization, if applicable). Informed consent processes and documentation must adhere to state laws/local requirements, including consent provided by the participant's legally authorized representative (LAR), responsible next of kin, surrogate consent with assent, etc.
2. Previously consented to participate in A3-45 screening.
3. Has A3-45 screening plasma biomarker results required for determining eligibility to participate in the A3-45 trial.
4. If an amyloid PET scan was conducted in A3-45, the scan was determined to be below the 20 centiloid cutpoint required for eligibility into the treatment arms of the A3 or A45 trial.
5. As assessed by the site PI, participant is likely to be able to comply with the protocol, including completion of all required procedures for the duration of the study, and has adequate vision, hearing (hearing aid permitted), and literacy in English or Spanish sufficient for compliance with required testing procedures.

Exclusion Criteria:

1. Current treatment with an FDA approved medication for Alzheimer's disease, including prior or current treatment with a prohibited medication.
2. Enrollment in another investigational study, or intake of investigational drug, within 30 days prior to screening, or five half-lives of the investigational drug, whichever is longer, unless it can be documented that the participant was in the placebo treatment arm.

   Participants enrolled in other observational studies may be permitted with Medical Monitor review and approval.
3. Screen failed from A3-45 due to not meeting basic inclusion criterion (i.e., age requirement; current diagnosis of AD dementia).

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll approximately 1000 participants who screen failed from the AHEAD study without evidence of elevated or intermediate amyloid by plasma biomarker or by amyloid PET scan at screening. Participants will have consented to participate in the AHEAD study and previously met demographic, cognitive and clinical criteria, however, had screening plasma biomarker and/or PET scan results that fell below the ABeta threshold levels required for randomization into the treatment arms for the AHEAD study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Rate of change from Baseline to Month 48 on plasma beta-amyloid (Aβ) 40 or 42 ratio | Baseline, Month 12, Month 24, Month 36 and Month 48
Rate of change from Baseline to Month 48 on plasma phosphorylated tau (ptau) 217 | Baseline, Month 12, Month 24, Month 36 and Month 48
  Assess longitudinal changes from initial visit in plasma phosphorylated tau (ptau) 217 ratio using a proteomics assay

SECONDARY OUTCOMES:
Rate of Change from Baseline to Month 48 as measured by the Preclinical Alzheimer Cognitive Composite 5(PACC5) | Baseline, Month 12, Month 24, Month 36 and Month 48
  PACC5:Free/cued selective reminding test:number of words recalled without cuing/with cuing(0[worst]-96[best recall]);Delayed Paragraph Recall test: recall of 1 short story(25 bits information),immediately after reading and again after delay of 30 minutes (0[worst]-25[best recall]);Digit-symbol substitution test: Participant uses a key to fill in blank squares as fast as possible in 90 seconds(0[none]-91[best performance]);Mini Mental State Score:to evaluate orientation, memory, attention, concentration, naming, repetition, comprehension and ability to create sentence, to copy 2 overlapping pentagons, scored as number of correctly completed items(0[worse]-30[perfect performance]);Category fluency task: participants generate words in 60 second belonging to a semantic category(total score:number of appropriate words generated per task, higher values indicate better performance).
Rate of Change from Baseline to Month 48 as measured Cognitive Function Index (CFI) | Baseline, Month 12, Month 24, Month 36 and Month 48
  CFI assessment to assess the participant's perceived ability to perform high-level functional tasks in daily life and sense of overall cognitive functional ability. Study participants (18 questions) and their study partners (15 questions) independently rate the participant's abilities. Total score combines participant and study partner scores, with higher scores indicating greater impairment. For participants, 0 = minimum;18 = maximum. For study partners, 0 = minimum; 15 = maximum. The CFI may be self-administered or completed as an interview conducted by clinical site personnel in-person or, if necessary, over the phone.

OTHER OUTCOMES:
Collection of baseline amyloid PET on participants without prior amyloid PET data | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul Aisen, MD, Study Director — University of Southern California (USC) Alzheimer's Therapeutic Research Institute (ATRI); Reisa Sperling, MD, Study Director — Brigham and Women's Hospital and Massachusetts General Hospital
Locations (56):
- United States (56):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California, Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Sharp Neurocognitive Research Center, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of California, Davis, Walnut Creek, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Brain Matters Research, Delray Beach, Florida
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - K2 Medical Research - The Villages, Lady Lake, Florida
  - K2 Medical Research, LLC, Maitland, Florida
  - Gonzalez MD & Aswad MD Health Services, Miami, Florida
  - Wien Center for Clinical Research, Miami Beach, Florida
  - Charter Research, Orlando, Florida
  - University of South Florida - Health Byrd Alzheimer Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas, Fairway, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Headlands Eastern MA LLC, Plymouth, Massachusetts
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University, St. Louis, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Las Vegas, Nevada
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Beachwood, Ohio
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Ohio, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Central States Research, LLC, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Butler Hospital Memory and Aging Program, Providence, Rhode Island
  - Ralph H. Johnson VA Health Care System, Charleston, South Carolina
  - Vanderbilt University Medical Center Center for Cognitive Medicine, Nashville, Tennessee
  - University of Texas, Southwestern MC at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Eastern Virginia Medical School at Old Dominion University, Norfolk, Virginia
  - National Clinical Research Inc., Richmond, Virginia
  - University of Washington, Memory and Brain Wellness Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- See also: Alzheimer's Clinical Trials Consortium — https://www.actcinfo.org/
- See also: Alzheimer's Therapeutic Research Institute — https://atri.usc.edu/
- See also: APEX Study Home Page — https://www.actcinfo.org/alzheimers-plasma-extension-apex-study/